CLINICAL TRIAL: NCT05385965
Title: Meaning-Centered Pain Coping Skills Training: A Randomized Controlled Trial of a Psychosocial Intervention for Advanced Cancer Patients
Brief Title: Meaning-Centered Pain Coping Skills Training for Cancer Pain
Acronym: MCPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00110762
Record Dates: First submitted 2022-04-27; First posted 2022-05-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Pain
Keywords: Caner pain management; Psychosocial intervention; Spiritual aspects of coping with pain; Pain Coping Skills Training; Meaning-Centered Psychotherapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned with equal allocation to an intervention or a standard care control condition, using a stratified block randomization scheme to ensure group balance based on patient performance status (i.e., Eastern Cooperative Oncology Group [ECOG] score of 0 vs. 1 or 2) and pain interference (i.e., Patient-Reported Outcomes Measurement Information System [PROMIS] Pain Interference 8-item raw score of 25 or lower vs. 26 or higher) at screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meaning-Centered Pain Coping Skills Training (Experimental): Four, 45-60 minute, videoconference-delivered sessions focus on training participants in cognitive and behavioral skills (e.g., guided imagery, activity pacing) for managing pain.
  Interventions: Behavioral: Meaning-Centered Pain Coping Skills Training
- Standard Care (No Intervention): Information and referrals for free services available through the Duke Cancer Patient Support Program.

INTERVENTIONS:
Behavioral: Meaning-Centered Pain Coping Skills Training — The goal of this intervention is to help participants reduce pain interference so that they can engage with what gives them a sense of meaning, purpose, and peace.
  Arms: Meaning-Centered Pain Coping Skills Training

SUMMARY:
This study is a randomized controlled trial of a psychosocial pain management intervention called, Meaning-Centered Pain Coping Skills Training (MCPC). Patients with advanced solid tumor cancer and pain interference (N=210) will be randomized to MCPC or a standard care control condition. Patient-reported outcomes will be assessed at baseline and 8- and 12-week follow-ups. The risk and safety issues in this trial are low and limited to those common to a psychosocial intervention (e.g., loss of confidentiality).

DETAILED DESCRIPTION:
Many patients with advanced cancer describe pain as a debilitating symptom that greatly interferes with activities they care about. Psychosocial interventions show promise for improving cancer-related pain; however, there is a lack of interventions that address existential and spiritual concerns (e.g., a loss of meaning, purpose, and peace) that are common among those facing high levels of pain interference from advanced cancer.

To address this need, an intervention called Meaning-Centered Pain Coping Skills Training (MCPC) was developed. In this trial, the investigators will randomize 210 patients to MCPC or enhanced usual care control. Patient-reported outcomes will be assessed at baseline and 8- and 12-weeks after baseline. As in the investigators' extensive pilot work, MCPC's four 45-to-60 minute individual weekly sessions will be delivered by trained study therapists via an accessible videoconference format. Intervention sessions focus on training participants in evidence-based cognitive-behavioral skills, such as guided imagery and activity pacing. Emphasis is placed on using skills to reduce the degree to which pain interferes with participants' sense of meaning, purpose, and peace.

The first aim of this trial is to determine the efficacy of MCPC for reducing the primary outcome of pain interference at 8-weeks. The second aim is to determine the efficacy of MCPC for improving secondary outcomes at 8-weeks. The third aim is to test the maintenance of MCPC's effects on primary and secondary outcomes at 12-weeks. The fourth aim is to estimate the cost-effectiveness of implementing MCPC.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV solid tumor cancer diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or lower
* At least one clinical pain severity rating > 0 out of 10 in past month
* At least moderate pain interference (8-item Patient-Reported Outcomes Measurement Information System [PROMIS] Pain Interference T-score >/= 55) in the past week at telephone screening
* Ability to speak and read in English
* Age >/= 18 years.

Exclusion Criteria:

* Significant cognitive impairment as indicated in medical chart or during telephone screening
* Serious untreated mental illness
* Primary brain cancer diagnosis
* Previous engagement in Pain Coping Skills Training or Meaning-Centered Psychotherapy
* Enrollment in hospice at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference-Short Form | 8-week follow-up
  This 8-item measure assesses the degree to which, over the past 7 days, pain has interfered with daily activities, work around the home, engagement in social activities, household chores, fun activities, enjoyment of social activities, enjoyment of life, and family life. Response options range from 1 (not at all) to 5 (very much). Higher scores indicate worse pain interference.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference-Short Form | 12-week follow-up
  This 8-item measure assesses the degree to which, over the past 7 days, pain has interfered with daily activities, work around the home, engagement in social activities, household chores, fun activities, enjoyment of social activities, enjoyment of life, and family life. Response options range from 1 (not at all) to 5 (very much). Higher scores indicate worse pain interference.
Brief Pain Inventory-Short Form (BPI-SF) Pain Severity Subscale | 8-week follow-up and 12-week follow-up
  This 4-item measure assesses pain severity at its worst, least, and average over the past 7 days as well as current pain severity. Response options range from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores indicate worse pain severity.
Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp) | 8-week follow-up and 12-week follow-up
  This 12-item measure references the past 7 days and includes an overall spiritual well-being score and three subscales: 1) meaning (i.e., reason for living, sense of meaning and purpose); 2) peace (i.e., feeling peaceful, sense of harmony within oneself); and 3) faith (i.e., finding strength and comfort in faith or spiritual beliefs). Response options range from 0 (not at all) to 4 (very much); two items are reverse coded. Higher scores indicate greater spiritual well-being.
Patient-Reported Outcomes Measurement Information System (PROMIS) Meaning and Purpose Scale | 8-week follow-up and 12-week follow-up
  This 8-item measure assesses feelings of meaning and purpose, including having a good sense of what makes one's life meaningful, a sense that one's life is valuable and worthwhile, having clear goals and aims, feeling life one's life has meaning, significance, direction, fulfillment, and purpose. Response options range from 1 (strongly disagree or not at all) to 5 (strongly agree or very much). Higher scores indicate greater meaning and purpose.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety-Short Form | 8-week follow-up and 12-week follow-up
  This 8-item measure assesses anxiety symptoms over the past 7 days, including fear, difficulty focusing on things other than anxiety, feeling overwhelmed by worries, feeling uneasy, nervousness, feeling the need for help with anxiety, feeling anxious, and feeling tense. Response options range from 1 (never) to 5 (always). Higher scores indicate worse anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression-Short Form | 8-week follow-up and 12-week follow-up
  This 8-item measure assesses depressive symptoms over the past 7 days, including feelings of worthlessness, helplessness, hopelessness, depression, failure, unhappiness, nothing to look forward to, and difficulty improving mood. Response options range from 1 (never) to 5 (always). Higher scores indicate worse depressive symptoms.
Chronic Pain Self-Efficacy Scale (CPS) | 8-week follow-up and 12-week follow-up
  This 5-item measures assesses patients' confidence regarding pain management, managing pain during daily activities, keeping pain from interfering with sleep, and confidence in their ability to reduce pain using methods other than taking additional medication. Response options range from 10 (not at all certain) to 100 (very certain). Higher scores indicate greater self-efficacy.
Medical Outcomes Study Social Support Survey (MOS-SS) | 8-week follow-up and 12-week follow-up
  This 8-item measure assesses how often someone was available to provide instrumental (i.e., practical) support and emotional support. Instrumental support includes having someone available if confided to bed, needing to visit a doctor, needing help preparing meals, and needing help with daily chores. Emotional support includes having someone available to have a good time with, turn to for suggestions, feel understood, and feel loved and wanted. Response options range from 1 (none of the time) to 5 (all of the time). Higher scores indicate greater social support.
5-item 5-level EuroQol Group (EQ-5D-5L) | 8-week follow-up and 12-week follow-up
  This 5-item measure assesses health-related quality of life across 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The response options range from 1 to 5, with response choices that vary per question. Higher scores indicate worse health-related quality of life.

OTHER OUTCOMES:
All-cause medical resource use | Baseline, 8-week follow-up, and 12-week follow-up
  Participants will report their medical resource use. This will include the number of hospitalizations and visits to the emergency department, urgent care, and outpatient clinics and current pain medication prescriptions. These variables will be collected for the past 30 days at baseline and since the previous time point at both follow-ups.
Participant time | 8-week follow-up
  The total number of minutes for each intervention session will be assessed.
Participant productivity | Baseline, 8-week follow-up, and 12-week follow-up
  Participants' will report the number of weekly hours they worked inside and outside of the home.
Therapist time | 8-week follow-up
  The total number of minutes that therapists spent preparing for, conducting, and documenting intervention sessions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G Winger, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No